CLINICAL TRIAL: NCT03240835
Title: The Function of Pre-Albumin, Retinol Conjugated Protein and Transferrin in Early Malnutrition Detecting and Nutritional Status Dynamic Monitoring for Local Advanced Nasopharyngeal Carcinoma Patients With Chemoradiotherapy
Brief Title: The Function of PA, RBP and TRSF in Malnutrition Detecting and Nutritional Status Monitoring for NPC Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhao Chong (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor-Investigator, Zhao Chong, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: NPC-PA/RBP/TRSF
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Nasopharyngeal Carcinoma; Malnutrition
Keywords: pre-Albumin; Retinol Conjugated Protein; Transferrin; Locoregionally Advanced Nasopharyngeal Carcinoma; nutrition
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Malnutrition | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCRT±NACT: Patients treated with neoadjuvant chemotherapy(NC) (cisplatin and docetaxel) and CCRT (cisplatin) , or treated with CCRT only
  Interventions: Drug: cisplatin and docetaxel; Radiation: IMRT

INTERVENTIONS:
Drug: cisplatin and docetaxel — NACt：cisplatin 75 mg/m2 intravenous infusion in day1，docetaxel 75 mg/m2 intravenous infusion in day1，both drugs are given every 3 weeks, two cycles.
  CCRT: cisplatin (100mg/m2 on day 1) every three weeks for two cycles.
Radiation: IMRT — intensity modulation radiation therapy

SUMMARY:
The purpose of this study is to study the function of pre-albumin, retinol conjugated protein and transferrin in early malnutrition detecting and nutritional status dynamic monitoring for local advanced nasopharyngeal carcinoma patients with chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal carcinoma(WHO II/III)
* All genders，range from 18～60 years old
* Karnofsky performance status(KPS) ≥ 80
* Clinical stage III~IVb(UICC 8th)
* Without significant digestive system disease，nutritional and metabolic diseases or endocrine disease
* Without significant cardiac，respiratory，kidney or liver disease
* Not received radiotherapy, chemotherapy and other anti-tumor treatment(including immunotherapy)
* white blood cell(WBC) count ≥ 4×109/L, neutrophile granulocyte(NE) count ≥ 1.5×109/L, Hemoglobin(HGB) ≥ 10g/L, platelet(PLT) count ≥ 100×109/L
* alanine aminotransferase (ALT) or aspartate aminotransferase(AST) < 1.5×upper limit of normal(ULN), bilirubin < 1.5×ULN, alanine aminotransferase (CCR) ≥ 30ml/min
* Inform consent form

Exclusion Criteria:

* Distance metastases
* Second malignancy within 5 years
* Drug or alcohol addition
* Do not have full capacity for civil acts
* Active systemic infections
* Chronic consumptions
* Mental disorder
* Pregnancy or lactation
* Concurrent immunotherapy or hormone therapy for other diseases
* Severe complication, eg, uncontrolled hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: III-IVb(Union for International Cancer Control,UICC 8th) NPC patients with histologic diagnosis of World Health Organization(WHO) II/III
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of PA/RBP/TRSF | baseline and during treatment
  to evaluate the changes of PA/RBP/TRSF during the treatment

SECONDARY OUTCOMES:
Change of Body weight | baseline and during treatment
  to compare the change of weight loss during treatment
Number of Participants With Abnormal Laboratory Values | baseline and during treatment
  To observe the complete blood cell count and blood biochemical examination during treatment
Acute Toxicity | baseline and during treatment
  To evaluate the acute toxicity with Common Terminology Criteria For Adverse Events (CTCAE) 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China